CLINICAL TRIAL: NCT07327996
Title: Evaluation of Post-operative Pain and Bacterial Load Reduction After Incorporation of Mesoporous Silica Nanoparticles in Calcium Hydroxide Intracanal Medicament in Mandibular First Molar Teeth With Necrotic Pulp. "Randomized Controlled Clinical Trial"
Brief Title: Evaluation of Pain Relief and Bacterial Reduction After Using Calcium Hydroxide With Mesoporous Silica Nanoparticles as an Intracanal Medicament in Necrotic Mandibular Molars: A Randomized Controlled Clinical Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Future University in Egypt (Other)
Responsible Party: Principal Investigator, raneem mohamed, principal investigator, Future University in Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: raneemICM10
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-10

CONDITIONS: Necrotic Pulp
Keywords: postoperative pain; bacterial load
MeSH Terms: conditions — Dental Pulp Necrosis; Pain, Postoperative | interventions — Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The root canals will be filled with calcium hydroxide paste (Active Comparator): using calcium hydroxide paste as intracanal medication for 1week
  Interventions: Procedure: Calcium Hydroxide Intracanal medication
- The root canal will be filled with mesoporous silica nanoparticles paste. (Active Comparator): using mesoporous silica nanoparticles paste as intracanal medication for week
  Interventions: Procedure: mesoporous silica nanoparticles paste
- root canals will be filled with mesoporous silica nanoparticles with calcium hydroxide paste. (Active Comparator): using mesoporous silica nanoparticles with calcium hydroxide paste as intracanal medication for 1week
  Interventions: Procedure: Calcium Hydroxide + mesoporous silica nanoparticles

INTERVENTIONS:
Procedure: Calcium Hydroxide Intracanal medication — root canals filled with calcium hydroxide paste as intracanal medication for 1week
  Arms: The root canals will be filled with calcium hydroxide paste
Procedure: mesoporous silica nanoparticles paste — root canals filled with mesoporous silica nanoparticles for 1 week
  Arms: The root canal will be filled with mesoporous silica nanoparticles paste.
Procedure: Calcium Hydroxide + mesoporous silica nanoparticles — Root canal filled with Intracanal medication by combination between mesoporous silica nanoparticles with calcium hydroxide paste for one week.
  Arms: root canals will be filled with mesoporous silica nanoparticles with calcium hydroxide paste.

SUMMARY:
This study compares how well different root canal medications reduce pain and bacteria after treatment of lower molar teeth with necrotic pulp. It tests whether adding mesoporous silica nanoparticles-antibacterial particles-to calcium hydroxide makes the treatment more effective. Forty-two adult patients will be randomly assigned to receive either calcium hydroxide alone, nanoparticles alone, or a mix of both for one week during root canal therapy. measure patients' pain levels after 6h,12h,24,48h and 72 hours from treatment and the number of bacteria before and after treatment to see which method gives the best results. The goal is to make root canal treatments more comfortable and successful for future patients.

ELIGIBILITY:
* Inclusion Criteria:

  1. Patients with an age range between 18 to 40.
  2. No sex predilection.
  3. Patients with necrotic pulp.
  4. Patients able to sign informed consent.
  5. Restorable teeth.
  6. Positive patient's acceptance for participating in the study.
  7. Type III distal and mesial canal of first mandibular molar.
* Exclusion Criteria:

  1. Pregnant females
  2. Medically compromised patients.
  3. Patients having analgesics before the treatment
  4. If antibiotics have been administrated during the past two weeks pre-operatively.
  5. Patients having bruxism or clenching
  6. Patients having sever malocclusion associated with traumatic occlusion.
  7. Teeth that have:

     1. Peri-apical radiolucency
     2. Root resorption.
     3. Pulp stones or calcifications.
     4. Previous endodontic treatment.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain after application of different intracanal medications | from 6 to 72 hours from the treatment
  measuring Post-operative pain by Numerical rate scale and pain level will be assigned to one of 4 categorical score: none(0) - mild(1-3), severe(7-10) after 6h,12h,24,48h

SECONDARY OUTCOMES:
bacterial load change after intracanal medication | immediately in the intervention and after 1 week
  Recording the percentage of bacterial load reduction by collecting samples by paper points, first sample after access cavity and before RCT, second sample after mechanical instrumentation, third sample after removing intracanal medication from the canal

CONTACTS AND LOCATIONS:
Locations (1):
- Future University in Egypt, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided